# BPIT\_2024\_Statistical Analysis Plan (SAP) – Version 1.0

**Protocol Title:** A Prospective, Single-Center, Interventional Study to Evaluate the 5-Line Principle of Balanced Intensity Training (BPIT) for Enhancing Physical Performance and

Reducing Injury Risk

Protocol ID: BPIT-GFFI-2024-001

ClinicalTrials.gov ID: WAITING (or the final NCT number once released)

SAP Version: 1.0

Date: 30 November 2024

Principal Investigator: Dr. Neeraj Mehta, PhD

Statistician: [Dr. Anupama Mahagan (PhD), Mathematics]

## 1. Objectives (directly from protocol)

## Primary

- To assess change from baseline to Week 6 in 1-repetition maximum (1RM) for squat, bench press, and deadlift
- To assess the incidence of training-related injuries over the 6-week period

# Secondary

- Change in resting heart rate and heart rate variability (HRV RMSSD)
- Change in heart rate recovery (HRR) if measured
- Change in muscle activation (EMG %MVC) for rectus abdominis and quadriceps
- Change in knee valgus angle and spinal curvature (degrees)

### 2. Analysis Populations

- Intention-to-Treat (ITT): All 23 enrolled participants
- Per-Protocol (PP): Participants with ≥80% session adherence (actual adherence was 94.9%, so PP ≈ ITT)
- Safety population: All participants who received at least one training session

### 3. Primary Efficacy Analysis

- Paired t-test (or Wilcoxon signed-rank test if normality violated) comparing baseline vs.
  Week 6 for each 1RM exercise
- Effect size: Cohen's d (paired)
- Summary: Mean ± SD at baseline and Week 6, mean change, 95% CI, p-value, Cohen's

# 4. Injury Incidence

- Proportion of participants with ≥1 training-related injury (with 95% Clopper-Pearson exact CI)
- Injury rate per 1,000 training hours

# 5. Secondary Efficacy Analyses

All continuous secondary endpoints analysed exactly as primary (paired t-test/Wilcoxon, Cohen's d, 95% CI)

# 6. Missing Data

No missing primary outcome data expected (all 23 participants completed the study). If any missing values occur, listwise deletion will be used (sensitivity analysis with last-observation-carried-forward if >5% missing).

# 7. Multiplicity

No adjustment for multiplicity is planned (exploratory single-arm study).

## 8. Interim Analysis

None planned.

### 9. Software

IBM SPSS 29 or R 4.4.x

# 10. Tables & Figures (to be produced)

Exactly the same tables and figures that already appear in your final report (Tables 2–5, Figures 1–4).

| Approved by: | |
|------------------------------------|------------------------|
| Dr. Neeraj Mehta (PI) | Date: 30 November 2024 |
| Dr. Anupama Mahajan (Statistician) | Date: 30 November 2024 |